CLINICAL TRIAL: NCT03691142
Title: A Retrospective Study of Obstetrical and Neonatal Complications in Hereditary Haemorrhagic Telangiectasia (HHT)
Brief Title: Evaluation of Obstetrical and Neonatal Complications in Hereditary Haemorrhagic Telangiectasia (HHT)
Acronym: CONCERTO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0267
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Osler Rendu Disease; Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Hereditary Haemorrhagic Telangiectasia: Women with Hereditary Haemorrhagic Telangiectasia with at least one full term pregnancy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Interview of women with Hereditary Haemorrhagic Telangiectasia (HHT) during a consultation in the Reference Center for HHT or through a phone questionnaire about obstetric history, complications during pregnancy, delivery and neonatal outcomes.

SUMMARY:
Hereditary Haemorrhagic Telangiectasia (HHT) is a rare inherited genetic disease of autosomal dominant inheritance with a prevalence of about 1/5000. It is manifested by haemorrhage, mucocutaneous telangiectasia and visceral arteriovenous malformations (AVMs) (lung, liver and nervous system).

Severe complications during pregnancy in HHT are rare but considered high risk. Intracranial or pulmonary haemorrhage, stroke and heart failure have been reported in some women with HHT during pregnancy. These complications occur most often in the second and third trimesters when maternal physiological changes such as peripheral vasodilatation and increased cardiac output are at their peak.

Previous retrospective studies were conducted with numbers ranging from 40 to 97 patients and highlighted the importance of early screening of complications and specific management.

The aim of this study is to describe, on a larger number of patients, the obstetric and neonatal complications in patients with HHT and followed in the French Reference Center for HHT.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years.
* Patients monitored for clinically confirmed Hereditary Haemorrhagic Telangiectasia (presence of at least three Curaçao criteria) and / or with molecular biology confirmation.
* Patients with at least 1 full term pregnancy between 1960 and 2018.
* Received information and no opposition to participate in the study.

Exclusion Criteria:

* No full term pregnancies.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with Hereditary Haemorrhagic Telangiectasia and one or more past pregnancies.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of complications during pregnancy | Interview time (about 15 minutes)
  The questionnaire consists in collecting obstetric history (number of pregnancies, abortions), complications during pregnancy, delivery type and neonatal outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence pour la maladie de Rendu-Osler Service Génétique Clinique Bâtiment A1 - Hôpital Femme-Mère-Enfant - Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No